CLINICAL TRIAL: NCT05691426
Title: Assessment of the Effect of Non-surgical Periodontal Treatment on Endothelial Function- a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Zahi BADRAN, Professor, University of Sharjah
Other Study IDs: REC-22-02-28-04-S
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Endothelial Dysfunction; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test: Periodontitis patients
  Interventions: Diagnostic Test: Assessment of pulse wave amplitude (PWA); Diagnostic Test: Salivary Nitric Oxide
- Control: Periodontally healthy patients
  Interventions: Diagnostic Test: Assessment of pulse wave amplitude (PWA); Diagnostic Test: Salivary Nitric Oxide

INTERVENTIONS:
Diagnostic Test: Assessment of pulse wave amplitude (PWA) — Assessment of pulse wave amplitude (PWA) through peripheral arterial tonometry (PAT) using the device EndoPAT (Itamar Medical)
Diagnostic Test: Salivary Nitric Oxide — assessment the levels of salivary Nitric Oxide using a Nitric Oxide colorimetric detection kit,

SUMMARY:
An association between periodontitis and endothelial dysfunction has been reported, suggesting that periodontitis presents an inflammatory burden to the cardiovascular system, that might lead to AVD. The study aims aim to assess whether non-surgical periodontal therapy enhances endothelial function in periodontitis patients using a non-invasive diagnostic device to assess endothelial function through PWA and the assessment of levels of salivary Endothelin-1, in a population of people in the UAE.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: periodontally healthy subjects.
* Group 2: patients with periodontitis stage III or IV and grades A,B or C.

Exclusion Criteria:

* Medical conditions: Diabetes,pregnancy,obesity,renal disease,patients with cardiovascular diseases including hypertension,recent myocardial infarction or unstable angina (within 3 months),congestive heart failure,valvular heart disease
* Heavy smokers(>10 cigarettes per day),
* Regular administration of drugs resulting in gingival hyperplasia,root planning in the past 6 months
* Regular administration of drugs resulting in gingival hyperplasia (such as cyclosporine and phenytoin)
* Recent antibiotic use (in the past 3 months)
* Non-surgical periodontal therapy in the past 6 monthsp

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the pool of patients consulting at Postgraduate teachingb clinics of the University Dental Hospital Sharjah
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
pulse wave amplitude | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Badran, Study Director — University of Sharjah
Locations (1):
- University Dental Hospital Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No